CLINICAL TRIAL: NCT00579839
Title: A Randomized Controlled Trial of Immediate Versus Delayed Cord Clamping in the Preterm Neonate
Brief Title: Trial of Immediate vs. Delayed Cord Clamping in the Preterm Neonate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CordClampingElimian
Record Dates: First submitted 2007-12-18; First posted 2007-12-24 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: PreTerm Birth; PreTerm Neonate
Keywords: PreTerm Birth; PreTerm Neonate; High risk pregnancy; Preterm Baby; Premature Baby; Cord Clamping; Milking the cord
MeSH Terms: conditions — Premature Birth | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Delayed Cord Clamping
  Interventions: Procedure: Delayed Cord Clamping
- B (Active Comparator): Immediate cord clamping
  Interventions: Procedure: Immediate Cord Clamping

INTERVENTIONS:
Procedure: Delayed Cord Clamping — Delayed Cord Clamping: 30-35 seconds after birth
  Arms: A
Procedure: Immediate Cord Clamping — Immediate Cord Clamping: within 5 seconds of birth
  Arms: B

SUMMARY:
To determine the short and long term effects of placental transfusion at birth by milking and delayed cord clamping of the umbilical cord in neonates born between 24 weeks 0 days and 34 weeks 0 days weeks' gestation.

DETAILED DESCRIPTION:
This study is intended to be a randomized controlled trial comparing immediate cord clamping which represents the current standard of care at Oklahoma University Medical Center with delayed cord clamping among preterm neonates born between 24 weeks and 34 weeks 0 days weeks' gestation. Allocation sequence will be generated by simple randomization using random number table in the stratum 24-28 weeks 6 days and 29 weeks to 34 weeks 0 days weeks' gestation stratum.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies
* Signed consent to participate in the trial

Exclusion Criteria:

* Major fetal anomaly or known fetal chromosomal abnormalities
* Multiple gestation
* Mothers with pregestational and gestational diabetes
* Refusal to participate in the trial

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2006-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To determine the short and long term effects of placental transfusion at birth by milking and delayed cord clamping of the umbilical cord in neonates born between 24 weeks 0 days and 34 weeks 0 days weeks' gestation. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Elimian, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Elimian A, Goodman J, Escobedo M, Nightingale L, Knudtson E, Williams M. Immediate compared with delayed cord clamping in the preterm neonate: a randomized controlled trial. Obstet Gynecol. 2014 Dec;124(6):1075-1079. doi: 10.1097/AOG.0000000000000556. PMID 25415157